CLINICAL TRIAL: NCT03478124
Title: The Role of the Neuropsychological Evaluation for Early Diagnosis of Progressive Supranuclear Palsy
Brief Title: Neuropsychological Evaluation for Early Diagnosis of PSP
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: NPsy-PSP
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Progressive Supranuclear Palsy; Cognitive Impairment
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSP patients: Patients suffering from Progressive Supranuclear Palsy (PSP)
  Interventions: Behavioral: Cognitive evaluation
- PD Patients: Patients suffering from Parkinson's disease (PD)
  Interventions: Behavioral: Cognitive evaluation

INTERVENTIONS:
Behavioral: Cognitive evaluation — An extensive battery of neuropsychological and motor tests was assessed: MMSE, FAB, MoCA, WCST, Stroop Test, TMT-A and B, Verbal fluency Test, ROCF copy and delayed recall, RAVLT, 6MWT, TUG, BBS.

SUMMARY:
The aim of this study is to better understand the nature of the cognitive decline in Progressive Supranuclear Palsy, the time of its development and the relation with the other cardinal features of the disease.

DETAILED DESCRIPTION:
Progressive Supranuclear Palsy (PSP) is a neurodegenerative disease characterized by vertical supranuclear gaze palsy, early balance dysfunction and falls. Tau-protein aggregation, mainly in the brainstem, is the disease hallmark. Because of the similarities with Parkinson's disease (PD), the diagnosis is made approximately 4 years after the symptoms onset. Cognitive deficits are a leading feature of PSP and they actually represent one of the four functional core domains in the revised diagnostic criteria. The aim of this study is to better understand the nature of this cognitive decline, the time of its development and the relation with the other cardinal features of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the criteria for idiopathic PD
* Patients fulfilling the criteria for PSP

Exclusion Criteria:

* Any other neurodegenerative disorders or medical conditions different from PD / PSP

Age Groups: Child, Adult, Older Adult
Study Population: 56 PSP patients (PSPp) and 56 PD patients (PDp) were enrolled and matched for sex, age and disease duration.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
MMSE | 1 year
  Mini-Mental State Examination
FAB | 1 year
  Frontal Assessment Battery
MoCA | 1 year
  Montreal Cognitive Assessment
WCST | 1 year
  Wisconsin Card Sorting Test
ST | 1 year
  Stroop Test
TMT-A and B | 1 year
  Trail Making Test Parts A & B
VFT | 1 year
  Verbal fluency Test
ROCF copy and delayed recall | 1 year
  Rey-Osterrieth complex figure test copy and delayed recall
RAVLT | 1 year
  Rey Auditory Verbal Learning Test

SECONDARY OUTCOMES:
6MWT | 1 year
  6 Minute Walk Test
TUG | 1 year
  Timed Up and Go Test
BBS | 1 year
  Berg Balance Scale

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's disease, Movement Disorders and Brain Injury Rehabilitation, "Moriggia-Pelascini" Hospital - Via Pelascini, 3, 22015, Gravedona ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: Undecided